CLINICAL TRIAL: NCT05240651
Title: Change in Stroke Volume Index After Diuresis for Patients With Decompensated Heart Failure
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-02048
Record Dates: First submitted 2022-02-13; First posted 2022-02-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Acute Decompensated Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective cohort study for 50 patients admitted to the cardiac care unit requiring clinically-indicated diuretic therapy for congestive heart failure. The purpose of this study is to assess the role of non-invasive cardiac output monitoring (NICOM) with the Starling Fluid Management System (Baxter Medical, Deerfield, IL) in determining volume status in patients with acute decompensated heart failure requiring intravenous diuretic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of congestive acute decompensated heart failure (preserved or reduced ejection fraction) requiring clinically indicated IV diuresis
2. Admission to coronary/cardiac intensive care unit or cardiac step down unit
3. Able to provide written informed consent
4. Anticipated need for IV diuretics > 24 hrs

Exclusion Criteria:

1. Prisoner, pregnancy or post-partum stage, or age < 18 years
2. Known allergy to sensory material or gel
3. End stage renal disease or need for CRRT
4. Inability or contraindication to do a passive leg raise with both extremities (i.e., balloon pump, impella, spinal injury, amputation)
5. Other situation that might increase subject risk, interfere with study procedures, or confound study findings based on the opinion of the clinician/investigator
6. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adults age > 18
  * Decompensated heart failure requiring clinically-indicated intravenous (IV) diuresis
  * Admission to the cardiac care unit (CCU) or the step down unit (SDU)
  * Ability to perform a passive leg raise (PLR)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Stroke Volume Index (SVI) after passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
  The Startling System non-invasive cardiac output monitoring (NICOM) device will use a proprietary algorithm to determine SVI. A passive leg raise (PLR) is then performed to increase preload and then the Starling System takes a second set of measurements to determine the parameters above as well as the change in stroke volume index.

SECONDARY OUTCOMES:
Change in Stroke Volume Index (SVI) before passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
  The Startling System non-invasive cardiac output monitoring (NICOM) device will use a proprietary algorithm to determine SVI. A passive leg raise (PLR) is then performed to increase preload and then the Starling System takes a second set of measurements to determine the parameters above as well as the change in stroke volume index.
Change in Stroke Volume Index (SVI) after passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
  The Startling System non-invasive cardiac output monitoring (NICOM) device will use a proprietary algorithm to determine SVI. A passive leg raise (PLR) is then performed to increase preload and then the Starling System takes a second set of measurements to determine the parameters above as well as the change in stroke volume index.
Change in estimated Cardiac Output (CO) before passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
  The Startling System non-invasive cardiac output monitoring (NICOM) device will use a proprietary algorithm to determine CO. A passive leg raise (PLR) is then performed to increase preload and then the Starling System takes a second set of measurements to determine the parameters above as well as the change in CO.
Change in estimated Cardiac Output (CO) after passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
  The Startling System non-invasive cardiac output monitoring (NICOM) device will use a proprietary algorithm to determine CO. A passive leg raise (PLR) is then performed to increase preload and then the Starling System takes a second set of measurements to determine the parameters above as well as the change in CO.
Change in estimated Cardiac Index (CI) before passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
  The Startling System non-invasive cardiac output monitoring (NICOM) device will use a proprietary algorithm to determine CI. A passive leg raise (PLR) is then performed to increase preload and then the Starling System takes a second set of measurements to determine the parameters above as well as the change in CI.
Change in estimated Cardiac Index (CI) after passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
  The Startling System non-invasive cardiac output monitoring (NICOM) device will use a proprietary algorithm to determine CI. A passive leg raise (PLR) is then performed to increase preload and then the Starling System takes a second set of measurements to determine the parameters above as well as the change in CI.
Change in heart rate before passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
Change in heart rate after passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
Change in Mean arterial pressure before passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)
Change in Mean arterial pressure after passive leg raise (PLR) | Baseline, At Discharge (up to 1 week)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Alviar, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to carlos.alviar@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.